CLINICAL TRIAL: NCT04467268
Title: Sleep Extension in Overweight Short Sleepers: A Randomised Controlled Trial:
Brief Title: Sleep Extension for Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: University Hospitals, Leicester (Other); University of Leicester (Other)
Responsible Party: Principal Investigator, Dr Iuliana Hartescu, Lecturer in Psychology, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LBO-SSEHS-SE_IH
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Short Sleep
Keywords: short sleep; insufficient sleep; sleep extension; diabetes risk
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Blood samples outcome assessor was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep extension intervention (Experimental): Intervention group participants met with an experienced sleep scientist to discuss and agree changes to their sleep and personal schedules. Discussions lasted 60-90 minutes, were informed by actigraphic sleep assessments from the baseline period, and aimed to increase TST by ≥1 hour/night. The structure and content of the "About Sleep", "Sleep Hygiene" and "Thoughts and Sleep" components of the online Sleepful application, a self-help sleep management programme. Advice was supported by the provision of self-help booklets addressing sleep hygiene and the management of pre-sleep cognitions which had been successfully trailed in an intervention for insomnia symptoms. Finally, to capitalize on the participant's motivation at recruitment, and optimize adherence, the newly agreed sleep schedule was written into an agreement which the participant was asked to sign, simulating a 'therapeutic contract'. Schedules were reviewed by telephone at the end of the first week and revised if required.
  Interventions: Behavioral: Sleep extension
- Control group (No Intervention): Participants in the control group were asked to continue with their habitual sleep schedule.

INTERVENTIONS:
Behavioral: Sleep extension — The sleep extension programme was designed around four alternative assumptions: 1) that among this group of habitual short sleepers, extending time in bed (TIB) would represent a significant behavioral change to established night-time and daytime routines; 2) that for practical purposes (accommodating personal, family and work schedules) extended time in bed is best anchored against typical rise-times; 3) that sleep onset may represent a particular challenge for those advancing habitual bed-times by over 1 hour each night; and 4) that in consenting to the trial, participants were motivated to make and sustain behavioral change.
  Arms: Sleep extension intervention

SUMMARY:
The study aims to examine the effects of a sleep extension intervention on the metabolic and cardio-vascular profile of obese people who present traditional diabetes risk factors, and who are habitually sleep deprived. Participants randomized to the intervention arm will complete a 6-week sleep extension intervention, whilst the control group will maintain their habitual sleep schedule. It is hypothesized that the sleep extension intervention will significantly increase total sleep time, and will be accompanied by significant metabolic-related changes.

DETAILED DESCRIPTION:
Recent epidemiological (survey) research, conducted in both in healthy populations and among those with existing chronic disease, shows that insufficient sleep can significantly contribute to ill health (including diabetes, heart disease and obesity). These findings have also been accompanied by credible explanatory mechanisms emphasising the role of sleep in regulating appetite, satiety, glucose and daytime stamina. Sleep extension, therefore, is a largely unexplored pathway for improving individual health, and reducing an existing risk of diabetes. If successful, increased sleep duration and quality could be adopted as an achievable public health intervention.

The study aims to recruit a total of 20 men, overweight, presenting traditional risks of developing diabetes, who are habitually short sleepers. Participants are then randomized, stratified by weight status, to a sleep extension group, or a control sleep monitoring group. Baseline measures include sleep actigraphy, continuous glucose monitoring, blood pressure, and a mixed-meal tolerance test; after the 6-week intervention, the same measures are repeated.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25 to 55 years (inclusive)
* Gender: Men
* BMI > 25kg/m2
* Average self-reported sleep duration of ≤ 6h per 24h
* Stable daily sleep/wake schedule
* Health risk screening score ≥ 2

Exclusion Criteria:

* Diagnosed sleep disorder as per DSM-5: e.g. insomnia, restless legs syndrome, moderate/severe Obstructive Sleep Apnoea; Epworth Sleepiness Score: <5
* Diagnosed chronic conditions, or medication, likely to interfere with regular sleep: T2D, chronic fatigue syndrome, fibromyalgia, COPD, uncontrolled depression/anxiety, other severe psychiatric illness, substance abuse.
* Night/evening shift work , regular time-zone travel, other circumstances preventing regular sleep schedule (e.g. very young children, carer at night for sick relatives etc)

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
Total sleep time (TST) | 24 hours
  Time asleep obtained every night, as measured by actigraphy (minutes).

SECONDARY OUTCOMES:
Time in Bed (TIB) | 24 hours
  Time between getting into and getting out of bed (minutes)
Sleep onset latency (SOL) | 24 hours
  Time to fall asleep (minutes)
Wake after sleep onset (WASO) | 24 hours
  Time awake after the first sleep period (minutes)
Glucose concentration | 3-hour mixed meal tolerance test blood plasma samples: prior to the test meal (0 minutes), and at 30, 60, 90, 120, 150, and 180 minutes
  Total area under the glucose concentration curve
Insulin concentration | 3-hour mixed meal tolerance test blood plasma samples: prior to the test meal (0 minutes), and at 30, 60, 90, 120, 150, and 180 minutes
  Total area under the insulin concentration curve
Total PYY concentration | 3-hour mixed meal tolerance test blood plasma samples: prior to the test meal (0 minutes), and at 30, 60, 90, 120, 150, and 180 minutes
  Total area under the PYY concentration curve
Grelin concentration | 3-hour mixed meal tolerance test blood plasma samples: prior to the test meal (0 minutes), and at 30, 60, 90, 120, 150, and 180 minutes
  Total area under the ghrelin concentration curve
Leptin concentration | 8-hour fasting blood samples
  Fasting leptin levels
Minutes per 24 hours of Moderate to vigorous physical activity (MVPA) | 24 hours
  Physical activity recorded with actigraphs
Standard Deviation of Blood Glucose Standard Deviation of Blood Glucose | 14 days
  Obtained from all CGMs 24-hour blood glucose concentrations across the monitoring period with
Mean Amplitude of Glycemic Excursions | 24 hours
  Mean blood glucose values exceeding one standard deviation of the 24-hour arithmetic average across the monitoring period
Systolic and diastolic blood pressure | 10 minutes
  Measurements of arterial blood pressure were taken, each after resting in a supine position for 10 minutes in a fasting state
Pittsburgh Sleep Quality Index | One month
  Self-reported measure of sleep quality, score range 0-21,higher scores indicate worse sleep quality.
Multidimensional Assessment of Fatigue | One week
  Self-reported assessment of experienced fatigue, scores range from 1 to 50, higher scores indicate worse fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Iuliana Hartescu, PhD, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hartescu I, Stensel DJ, Thackray AE, King JA, Dorling JL, Rogers EN, Hall AP, Brady EM, Davies MJ, Yates T, Morgan K. Sleep extension and metabolic health in male overweight/obese short sleepers: A randomised controlled trial. J Sleep Res. 2022 Apr;31(2):e13469. doi: 10.1111/jsr.13469. Epub 2021 Aug 29. PMID 34459060